CLINICAL TRIAL: NCT04643548
Title: Neurological Abnormalities in SARS-CoV-2 ICU Patients. A Prospective Study. NeuroCOVID Study
Brief Title: WHO Covid 19 - Neurological Abnormalities in SARS-CoV-2 ICU Patients
Acronym: NeuroCovid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: NeuroCovid-RNI 2020 GODET
Record Dates: First submitted 2020-11-16; First posted 2020-11-25 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: SARS-CoV-2 Infection; Intensive Care Unit Patient; Neurological Abnormality; Delirium; Encephalopathy
Keywords: SARS-CoV-2 infection; Intensive care unit patient; Neurological abnormalities; Delirium; Encephalopathy
MeSH Terms: conditions — COVID-19; Nervous System Malformations; Delirium; Brain Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The SARS-CoV-2 epidemic is leading to a large number of patients in intensive care units due to severe hypoxemic pneumonia. After an acute phase that may require controlled mechanical ventilation and deep sedation, removal of sedation often reveals a pathological awakening in the vast majority of patients. This encephalopathy state remains, to date and to our knowledge, unexplained. Clinical features do not appear to fully correlate with regular delirium. This encephalopathy might be explained by deep and prolonged hypoxemia, a wide use of sedation drugs, systemic inflammation or the hostile ICU environment.

DETAILED DESCRIPTION:
This study is intended to investigate neurological abnormalities associated with SARS-CoV-2 infection. Complete daily neurological examinations will be routinely conducted in intensive care unit patients. Specific biological analyses will also be performed in these patients by collecting additional blood samples from an arterial or central catheter, every 2 days. These clinical and biological examinations will be continued throughout patient's stay in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* COVID-19 positive patient (positive RT PCR, nasopharyngeal or tracheal)
* Patient admitted in an intensive care unit of the department of Anesthesia, Critical Care and Perioperative of Clermont-Ferrand University Hospital
* Patient with an arterial or central catheter to perform blood samples collection

Exclusion Criteria:

* Patient or family member's refusal to participate
* Neuropsychiatric history that may interfere with neurological evaluations in the intensive care unit
* Patient not affiliated with French social security insurance
* Patient under legal guardianship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in Intensive Care Unit and infected bye SARS-CoV-2
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-06-13 (Estimated); Study Completion 2021-08-13 (Estimated)

PRIMARY OUTCOMES:
Dosage of biomarkers typically explored in intensive care unit delirium | Change from Day 0 (= First day in ICU) until the end of the stay (up to 3 months) - Assessments every 2 days
  Plasminogen activator inhibitor-1 (PAI-1), E-selectin and angiopoietin-2
Dosage of neuronal injury markers | Change from Day 0 (= First day in ICU) until the end of the stay (up to 3 months) - Assessments every 2 days
  S100 β, Neuron Specific Enolase (NSE), GFAP, UCHL1, NFL

SECONDARY OUTCOMES:
Delirium assessment | Change from Day 0 (= First day in ICU) until the end of the stay (up to 3 months) - Assessments every days
  CAM-ICU (Confusion Assessment Method - Intensive Care Unit) scale
Delirium assessment | Change from Day 0 (= First day in ICU) until the end of the stay (up to 3 months) - Assessments every days
  ICDSC (Intensive Care Delirium Screening Checklist) scale.
Coma assessment | Change from Day 0 (= First day in ICU) until the end of the stay (up to 3 months) - Assessments every days
  CRS-R (Coma Recovery Scale-Revised)
Pupils characteristics | Change from Day 0 (= First day in ICU) until the end of the stay (up to 3 months) - Assessments every days
  Clinical observation
Pupils characteristics | Change from Day 0 (= First day in ICU) until the end of the stay (up to 3 months) - Assessments every days
  Pupilometer assessment
Neurological abnormalities | Change from Day 0 (= First day in ICU) until the end of the stay (up to 3 months) - Assessments every days
  Electroencephalogram : epileptic activity (spikes, spike-waves) or encephalopathy activity (triphasic waves))
Neurological abnormalities | Change from Day 0 (= First day in ICU) until the end of the stay (up to 3 months) - Assessments every days
  CT-scan
Neurological abnormalities | Change from Day 0 (= First day in ICU) until the end of the stay (up to 3 months) - Assessments every days
  MRI

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: Undecided